CLINICAL TRIAL: NCT06489574
Title: A Comparison Between Dexmedetomidine and Fentanyl as Adjuvants to Thoracic Epidural in Patients Undergoing Thoracotomy Surgery: A Randomized Controlled Trial
Brief Title: Dexmedetomidine and Fentanyl as Adjuvants to Thoracic Epidural
Acronym: adjuvants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed gamal solimn, director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD-249-2022
Record Dates: First submitted 2023-09-22; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Post-operative Pain; Thoracic Epidural; Thoracotomy Surgery
Keywords: Thoracotomy; Dexmedetomidine; Thoracic Epidural; Fentanyl
MeSH Terms: conditions — Pain, Postoperative | interventions — Tea; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized using a computer-generated list of random numbers, which will be sealed in closed envelopes. Patients will be randomly allocated to one of two groups; Group I will receive dexmedetomidine, while Group II (R) will receive fentanyl. An anesthesiologist who is not involved in the data collection team will perform all thoracic epidural infusion. Intra- and postoperative data will be collected by an anesthesiologist or intensivist who is blinded to the study protocol. So, both the patients and data collector were blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thoracic epidural with dexmedetomidine (Experimental): Patients will receive 50 μg dexmedetomidine with 10 ml of 0.125% bupivacaine followed by a continuous infusion of (10 ml bupivacaine + 25 μg dexmedetomidine + 39 ml saline with rate of 5 ml per hour)
  Interventions: Procedure: thoracic epidural with dexmedetomidine in patients undergoing thoracotomy surgery
- thoracic epidural with fentanyl (Experimental): Patients will receive 50 μg fentanyl in addition to 10 ml 0.125% bupivacaine followed by a continuous infusion (10 ml bupivacaine + 100 μg fentanyl + 38 ml saline with rate of 5 ml per hour)
  Interventions: Procedure: thoracic epidural with fentanyl in patients undergoing thoracotomy surgery

INTERVENTIONS:
Procedure: thoracic epidural with dexmedetomidine in patients undergoing thoracotomy surgery — A thoracic epidural catheter will be inserted at the T6- T7 intervertebral space, with the patient in the sitting position with standard aseptic precautions using an 18-G Touhy needle via a midline or paramedian approach with a loss of resistance method. A test dose of 3 ml of 2% lignocaine with adrenaline 5 µ/ml will be administered.
  For thoracic surgery the sensory dermatome blockade needs to cover the incision and intercostal drains and may extend from T4 to T8.
  The epidural drug will be administered according to the group allocation over a period of 10 minutes as follows:
  Group A:
  Patients will receive 50 μg dexmedetomidine with 10 ml of 0.125% bupivacaine followed by a continuous infusion of (10 ml bupivacaine + 25 μg dexmedetomidine + 39 ml saline with rate of 5 ml per hour).
  Arms: thoracic epidural with dexmedetomidine
Procedure: thoracic epidural with fentanyl in patients undergoing thoracotomy surgery — A thoracic epidural catheter will be inserted at the T6- T7 intervertebral space, with the patient in the sitting position with standard aseptic precautions using an 18-G Touhy needle via a midline or paramedian approach with a loss of resistance method. A test dose of 3 ml of 2% lignocaine with adrenaline 5 µ/ml will be administered.
  For thoracic surgery the sensory dermatome blockade needs to cover the incision and intercostal drains and may extend from T4 to T8.
  The epidural drug will be administered according to the group allocation over a period of 10 minutes as follows:
  Group B:
  Patients will receive 50 μg fentanyl in addition to 10 ml 0.125% bupivacaine followed by a continuous infusion (10 ml bupivacaine + 100 μg fentanyl + 38 ml saline with rate of 5 ml per hour).
  Arms: thoracic epidural with fentanyl

SUMMARY:
To find out if there is a benefit from adding dexmedetomidine to epidural bupivacaine as regards:

* Intra and postoperative opioid consumption
* Pain score (numerical rating scale)
* Hemodynamic stability,
* Patient satisfaction.

DETAILED DESCRIPTION:
Following approval from Research Committee of Anesthesia Department and the Ethics Committee of the Faculty of Medicine, Cairo University, 50 patients will be included in the study (25 patients per group). After obtaining written informed consents, all patients will be subjected to systematic preoperative assessment including history taking, physical examination, and review of the results of routine investigations. Upon arrival to the preparation room, a 20G IV cannula will be inserted into a peripheral vein and midazolam 2-3 mg will be administered unless contraindicated. A 20G arterial catheter will be inserted into the radial artery of the dependent (non-operative) side, after local infiltration with lidocaine 2%. Patients will be transferred to the operating room where routine monitoring is applied, including electrocardiography (ECG), invasive Blood Pressure (IBP) and pulse oximetry are attached. Baseline heart rate, blood pressure, oxygen saturation and respiratory rate will be recorded.

A thoracic epidural catheter will be inserted at the T6- T7 intervertebral space, with the patient in the sitting position with standard aseptic precautions using an 18-G Touhy needle via a midline or paramedian approach with a loss of resistance method. A test dose of 3 ml of 2% lignocaine with adrenaline 5 µ/ml will be administered.

For thoracic surgery the sensory dermatome blockade needs to cover the incision and intercostal drains and may extend from T4 to T8.

The epidural drug will be administered according to the group allocation over a period of 10 minutes as follows:

Group A:

Patients will receive 50 μg dexmedetomidine with 10 ml of 0.125% bupivacaine followed by a continuous infusion of (10 ml bupivacaine + 25 μg dexmedetomidine + 39 ml saline with rate of 5 ml per hour).

Group B:

Patients will receive 50 μg fentanyl in addition to 10 ml 0.125% bupivacaine followed by a continuous infusion (10 ml bupivacaine + 100 μg fentanyl + 38 ml saline with rate of 5 ml per hour).

After documenting the sensory blockade by using a piece of ice or cold object, If sensory level fail to be achieved, patient will be out of the study. Anesthesia will be induced with Propofol 2-3 mg/kg, together with fentanyl 2 mg/kg until loss of verbal response. Muscle relaxation will be achieved with atracurium 0.5 mg/kg and the patient's trachea will be intubated using a single or double-lumen tube, as indicated by the surgical procedure. Anesthesia will be maintained by isoflurane, and muscle relaxation will be maintained with atracurium 0.3 - 0.5 mg/kg/hr.

The lungs will be ventilated with positive pressure ventilation to maintain end-tidal carbon dioxide (EtCO2) between 32 and 36 mmHg.

Patients' heart rate, blood pressure will be monitored continuously and recorded at ten-minute intervals until the end of surgery. Any attack of hypotension, defined as a drop of > 20% of baseline blood pressure, will be managed by ephedrine 0.2 mg/kg IV, and administering I.V. fluids. On the other hand, hypertension, defined as an increase of > 20 % of baseline blood pressure, will be managed by increasing the depth of anesthesia and administering bolus doses of fentanyl 1 mic/kg (up to 3 mic/kg maximum dose).

Bradycardia (heart rate < 50 beats/min) will be managed by atropine 0.02 mg/ kg IV

At the end of surgery residual neuromuscular blockade will be reversed and the endotracheal tube will be removed. Patients will be transferred to the ICU and will be monitored for 24 hours. Patients' heart rate, blood pressure, oxygen saturation and respiratory rate will be monitored at regular intervals and the pain score and sedation level as well.

Epidural infusion will be continued with the same infusion rate. A fixed dose of paracetamol (10 - 15 mg/kg) every 8 hours and NASID (0.5 - 2/kg/ day divided in 2 doses will be administered I.V.

Pain will be assessed using the numerical rating scale (NRS) and if the pain score is more than 3, 3mg morphine I.V. will be administrated intra venous as rescue analgesia (up to .4 mg/kg morphine maximum dose every 24 Hours).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years old
* ASA physical status I-II-III
* Good mental function.
* Patient scheduled for thoracic surgery with posterolateral thoracotomy.
* BMI of patient (18 - 30).

Exclusion Criteria:

* Age less than 18 or more than 60 years old
* Any contraindications to epidural injection (patient refusal, local infection at the site of injection, coagulopathy, patients on anticoagulant or antiplatelet drugs, known allergy to local anesthetics, significant spine deformity)
* Inability to provide informed consent or pain score

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Total amount of morphine consumption in milligram in the first 24-hour postoperative in the two groups | 24 hours
  Dexmedetomidine compared to fentanyl as adjvant for thoracic epidural for post operative analgesia

SECONDARY OUTCOMES:
Systolic arterial blood pressure in millimetre mercury | Intraoperative
  will be recorded at baseline, ten and twenty minutes after epidural activation, immediately after induction, and every 10 minutes till end of surgery
heart rate (beat/ minute) | Intraoperative
  will be recorded at baseline, ten and twenty minutes after epidural activation, immediately after induction, and every 10 minutes till end of surgery
Diastolic arterial blood pressure in millimetre mercury | Intraoperative
  will be recorded at baseline, ten and twenty minutes after epidural activation, immediately after induction, and every 10 minutes till end of surgery
mean blood pressure n millimetre mercury | Intraoperative
  will be recorded at baseline, ten and twenty minutes after epidural activation, immediately after induction, and every 10 minutes till end of surgery
Pain Score According to Numerical Rating Scale (NRS) | 24 Hours
  The pain score will be assessed using the NRS, where patients will rate their pain on a scale from 0 to 10. The NRS value will be obtained from the patient immediately after recovery from anesthesia and then every 4 hours during the first 24 hours postoperatively.
  Minimum Value: 0 (no pain) Maximum Value: 10 (worst possible pain) Interpretation: Higher scores indicate worse outcomes (more severe pain).
First request of analgesia postoperative | 24 Hours post operative
  The elapsed time from the start of thoracic epidural infusion until the administration of the first postoperative rescue analgesia in hours
Patient Satisfaction with Epidural Infusion | 24 hours
  Patient satisfaction will be assessed using a validated satisfaction survey immediately after the procedure. The survey will include questions rated on a Likert scale from 1 to 5, where 1 indicates "very dissatisfied" and 5 indicates "very satisfied." Minimum Value: 1 (very dissatisfied) Maximum Value: 5 (very satisfied) Interpretation: Higher scores indicate greater satisfaction with the procedure
Incidence of side effects | 24 hours
  (nausea, vomiting, shivering, hypotension, dizziness, dry mouth, and respiratory depression)

CONTACTS AND LOCATIONS:
Overall Officials: mohamed g soliman, MS, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Wenk M, Schug SA. Perioperative pain management after thoracotomy. Curr Opin Anaesthesiol. 2011 Feb;24(1):8-12. doi: 10.1097/ACO.0b013e3283414175. PMID 21084984
- [Background] Salomaki TE, Laitinen JO, Nuutinen LS. A randomized double-blind comparison of epidural versus intravenous fentanyl infusion for analgesia after thoracotomy. Anesthesiology. 1991 Nov;75(5):790-5. doi: 10.1097/00000542-199111000-00010. PMID 1952204
- [Background] Amr YM, Yousef AA, Alzeftawy AE, Messbah WI, Saber AM. Effect of preincisional epidural fentanyl and bupivacaine on postthoracotomy pain and pulmonary function. Ann Thorac Surg. 2010 Feb;89(2):381-5. doi: 10.1016/j.athoracsur.2009.10.060. PMID 20103303
- [Background] Shaikh SI, Mahesh SB. The efficacy and safety of epidural dexmedetomidine and clonidine with bupivacaine in patients undergoing lower limb orthopedic surgeries. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):203-9. doi: 10.4103/0970-9185.182104. PMID 27275050
- [Background] Sathyanarayana LA, Heggeri VM, Simha PP, Narasimaiah S, Narasimaiah M, Subbarao BK. Comparison of Epidural Bupivacaine, Levobupivacaine and Dexmedetomidine in Patients Undergoing Vascular Surgery. J Clin Diagn Res. 2016 Jan;10(1):UC13-7. doi: 10.7860/JCDR/2016/17344.7079. Epub 2016 Jan 1. PMID 26894153
- [Background] Karhade SS, Acharya SA, Harnagale K. Comparative analysis of epidural bupivacaine versus bupivacaine with dexmedetomidine for vaginal hysterectomy. Anesth Essays Res. 2015 Sep-Dec;9(3):310-3. doi: 10.4103/0259-1162.158007. PMID 26712965
- [Background] Bajwa SJ, Arora V, Kaur J, Singh A, Parmar SS. Comparative evaluation of dexmedetomidine and fentanyl for epidural analgesia in lower limb orthopedic surgeries. Saudi J Anaesth. 2011 Oct;5(4):365-70. doi: 10.4103/1658-354X.87264. PMID 22144922
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT06489574/Prot_SAP_000.pdf